CLINICAL TRIAL: NCT04233307
Title: Non-invasive Assessment of Perfusion and the Risk of Wound Complication in High Risk Surgical Incisions
Brief Title: Wound Perfusion in High Risk Surgical Incisions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Florida Orthopaedic Institute (Network)
Responsible Party: Principal Investigator, Barbara Steverson, Director of Research, Orthopaedic Trauma Service, Florida Orthopaedic Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: USF000305
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Bone Fractures Multiple
Keywords: perfusion
MeSH Terms: conditions — Fractures, Multiple

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wound photographs (Other): Telethermographic photographs of fracture wound and contralateral limb before and after propofol infusion.
  Interventions: Diagnostic Test: Telethermographic images

INTERVENTIONS:
Diagnostic Test: Telethermographic images — Infrared digital thermography photographs of fracture wound and contralateral limb before and after propofol infusion.
  Other Names: Forward-Looking Infrared (FLIR) photographs

SUMMARY:
This is a prospective cohort pilot study. The primary purpose is to report the perfusion status of the surgical field in at risk surgical incisions. The secondary purposes are to describe the relationship between perfusion status and wound healing status and complications, and to describe the relationship between infrared digital thermography perfusion readings and the timing of propofol infusion. The research intervention will be photographs taken of the wound on the injured extremity, with a Forward-Looking Infrared (FLIR) camera, for the purpose of assessing perfusion status and skin temperature at the surgical site.

DETAILED DESCRIPTION:
Patients with qualifying injuries will be identified at the time of injury. There will be no deviation from standard of care for these patients outside of the acquisition of the FLIR image. Standard emergent management of these injuries including but not limited to reduction, immobilization, and acquisition of advanced imaging will take place. Pre-operative discussion of the risks and benefits of surgical management will occur and informed consent obtained.

Propofol is a commonly used anesthetic agent. However, propofol is also a vasodilating agent, which acts by blocking sympathetic tone. Limited worked has been done to evaluate the effects of propofol administration on the FLIR imaging data acquisition. A single study used FLIR to look at tissue perfusion after propofol infusion in children. In this study, the primary concern was whether infrared imaging could replace or augment, serial blood pressure and heart rate measurements, or other invasive monitoring measurements in patients undergoing general anesthesia with the use of vasodilatory agents, such as propofol. The authors' goal was to "assess the ability of the thermal imager to trend heat loss that registers as skin temperature from propofol-mediated vasodilation and study reversibility as propofol levels drop and vascular tone returns." This leaves a void regarding surgeons' understanding of the optimal timing of FLIR perfusion assessment and the reliability of measurements obtained pre and post propofol infusion.

In order to better understand the effects of propofol and determine the optimal time for determining perfusion with the FLIR camera, the investigators will take a first reading in the pre-operative holding area, prior to the administration of any propofol or other vaso-active agent (as described below). Once in the operating room, after the induction of anesthesia but prior to application of any topical cleansing or cooling products to the skin, the participant will be transferred to the operating room table and placed on a clean, white sheet and blankets will be removed from both lower extremities. The planned surgical incision(s) to be used will be drawn on the skin by the most senior surgeon. Next, a clinical photo and a FLIR image will be obtained at 90 degrees to the skin, and 1 meter from the surface of the skin at the site of each planned incision. One researcher has successfully used a protocol of taking images at perpendicular to the skin and 1 meter distance and demonstrated that deviation of as much as 20 degrees from the perpendicular and 0.5m of distance has negligible effect on readings. A set of control photos, identical to the ones obtained on the injured extremity will be obtained on the contralateral, non-injured extremity. A physician who is part of the surgical team who is trained in the use of the FLIR camera will obtain the images. At the time of image acquisition, results of the wrinkle test at each incision, patient body temperature, room temperature and humidity will be recorded. Analysis of the FLIR images will involve averaging the tissue perfusion in a box drawn with 1 cm borders around the planned incision site as well as the entire area imaged. This will be compared to the control, the contralateral uninjured extremity.

Participants will receive standard operative management of these injuries with standard of care post-operative management.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patients, with talus, calcaneus, tibial plafond, trimalleolar ankle fracture-dislocations, lisfranc, or tibial plateau fractures who are indicated for surgical management in the form of open reduction and internal fixation or external fixation.

Exclusion Criteria:

1. Pathologic Fracture
2. Previous open surgery in the operative field
3. Prisoners
4. Systemic skin disorder affecting the surgical field
5. Vascular Injury involving vessel that supplies the surgical field
6. Bilateral qualifying lower extremity injuries
7. Homeless
8. Those unable to follow up through the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Soft tissue healing | 2 weeks post-operative
  The number of patients with the expected level of incision healing appropriate to the time frame per Clinician judgement
Soft tissue healing | 6 weeks post-operative
  The number of patients with the expected level of incision healing appropriate to the time frame per Clinician judgement
Soft tissue healing | 3 months post-operative
  The number of patients with the expected level of incision healing appropriate to the time frame per Clinician judgement
Soft tissue healing | 6 months post-operative
  The number of patients with the expected level of incision healing appropriate to the time frame per Clinician judgement

SECONDARY OUTCOMES:
Additional wound care intervention needed | within the 2 week post-operative period
  The number of participants requiring topical wound care, oral antibiotics, repeat surgical debridement, soft tissue coverage procedure or amputation required
Additional wound care intervention needed | within the 6 week post-operative period
  The number of participants requiring topical wound care, oral antibiotics, repeat surgical debridement, soft tissue coverage procedure or amputation required
Additional wound care intervention needed | within the 3 month post-operative period
  The number of participants requiring topical wound care, oral antibiotics, repeat surgical debridement, soft tissue coverage procedure or amputation required
Additional wound care intervention needed | within the 6 month post-operative period
  The number of participants requiring topical wound care, oral antibiotics, repeat surgical debridement, soft tissue coverage procedure or amputation required

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Mir, MD, Principal Investigator — Florida Orthopaedic Institute

IPD SHARING:
Plan to Share IPD: No